CLINICAL TRIAL: NCT07071142
Title: Frailty and 6-Month Clinical Outcomes in Elderly Patients With Heart Failure and Left Ventricular Ejection Fraction >40%
Brief Title: Frailty and Outcomes in Older Heart Failure Patients With Ejection Fraction >40%
Status: Active, not recruiting | Type: Observational
Sponsor: Duyen Nguyen Hoang Mai (Other)
Responsible Party: Sponsor-Investigator, Duyen Nguyen Hoang Mai, Resident Physician, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Other Study IDs: NT62722030
Record Dates: First submitted 2025-07-07; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Frailty Syndrome; Heart Failure and Mildly Reduced Ejection Fraction; Heart Failure and Preserved Ejection Fraction
Keywords: frailty; heart failure; Elderly; outcome; outpatient; age over 60; EF>40%; ejection fraction above 40%
MeSH Terms: conditions — Frailty; Heart Failure; Heart Failure, Diastolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the prevalence of frailty and its association with six-month clinical outcomes in elderly patients with heart failure and left ventricular ejection fraction greater than 40%. Elderly patients diagnosed with heart failure will be assessed for frailty status and followed up for six months to evaluate outcomes such as hospitalization and mortality. The study is observational and will help improve understanding of the impact of frailty on the prognosis of heart failure patients with ejection fraction >40%.

DETAILED DESCRIPTION:
This observational cohort study aims to evaluate the prevalence of frailty and its association with six-month clinical outcomes, including hospitalization and mortality, in elderly patients with heart failure (HF) and left ventricular ejection fraction (LVEF) >40%.

The study is conducted at the Cardiology outpatient clinics of Thong Nhat Hospital and the Heart Failure Clinic of the University Medical Center, Ho Chi Minh City, Vietnam. A total of approximately 301 patients aged ≥60 years with HF and LVEF >40% (per ESC 2021 criteria) will be enrolled. Baseline assessments include demographic and clinical characteristics, geriatric syndromes, and laboratory findings. Frailty will be assessed using Fried criteria; functional status using Katz ADL and Lawton IADL; nutritional status using the Mini Nutritional Assessment (MNA); depression using the Geriatric Depression Scale-15 (GDS-15); and polypharmacy, comorbidities, and falls will also be recorded.

Participants will be followed for six months to collect data on hospitalizations, mortality, and other adverse clinical outcomes. Data collection will be performed by trained investigators using standardized case report forms (CRFs) and entered into a secure electronic database. Data will undergo regular quality checks for accuracy, completeness, and consistency, with predefined range and logic checks, and source data verification against medical records for a random sample of participants.

Standard Operating Procedures (SOPs) are implemented to ensure uniformity in patient recruitment, informed consent, data collection, follow-up, and adverse event reporting. A data dictionary describing all variables, coding schemes, and normal reference ranges has been developed and will be maintained. Missing data will be documented and addressed using appropriate imputation or sensitivity analyses as outlined in the statistical analysis plan (SAP).

The sample size of approximately 301 participants is based on an expected frailty prevalence of ~50% in this population, allowing estimation with acceptable precision and adequate power to detect associations with outcomes. Statistical analyses will include descriptive statistics, Kaplan-Meier survival analysis, and multivariable regression modeling to assess the relationship between frailty and clinical outcomes while adjusting for potential confounders.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of heart failure with left ventricular ejection fraction >40% (per ESC 2021 guidelines).
* Attending outpatient cardiology clinics at Thong Nhat Hospital or Heart Failure Clinic at University Medical Center, Ho Chi Minh City during the study period.
* Vietnamese nationality.
* Able to communicate or have a caregiver who understands the patient's condition.
* Willing and able to provide informed consent.

Exclusion Criteria:

* Terminal illness with life expectancy <6 months due to other causes as assessed by the investigator.
* Severe dementia or severe mental illness preventing accurate interview or follow-up.
* Severe visual or hearing impairment affecting data collection.
* Unable to provide reliable medical history.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly patients (≥60 years) with heart failure and left ventricular ejection fraction >40%, attending the cardiology outpatient clinics at Thong Nhat Hospital and the Heart Failure Clinic at University Medical Center, Ho Chi Minh City, Vietnam, during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 301 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Composite of All-Cause Mortality or Hospitalization | 6 months after enrollment
  The number of participants who experience any of the following within 6 months after enrollment: all-cause mortality, cardiovascular mortality, all-cause hospitalization, or hospitalization for heart failure. The composite outcome includes either death or hospitalization from any cause. Events are verified from medical records and caregiver interviews.

CONTACTS AND LOCATIONS:
Locations (2):
- Vietnam (2):
  - Thong Nhat Hospital - Cardiology Outpatient Clinic, Ho Chi Minh City, Ho Chi Minh
  - University Medical Center Ho Chi Minh City - Heart Failure Clinic, Ho Chi Minh City, Ho Chi Minh

IPD SHARING:
Plan to Share IPD: No
Information Security